CLINICAL TRIAL: NCT04013503
Title: National Tunisian Registry of Hypertension
Acronym: NATURE-HTN
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: DAC-006-NATUREHTN
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
Keywords: NATURE-HTN
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Tunisian Society of Cardiology and Cardiovascular Surgery (STCCCV) proposes to coordinate a national, observational, cross-sectional and multicenter survey carried out during one month. The main objective of the survey is to describe the blood pressure and cardiovascular risk profile of the hypertensive patient in Tunisia.

This survey will allow us to have a generalized and updated view of the tunisian hypertensive patient in order to optimize treatment and to know the degree of adherence of practitioners to international recommendations in the care of the hypertension in Tunisia.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Informed consent, read and signed

Exclusion Criteria:

Consent not obtained

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting in consultation of cardiology, general medicine / family medicine, internal medicine and nephrology will be recruited in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Level | At inclusion
  Mean of Systolic and Diastolic Blood Pressure in mmHg
Cardiovascular Risk Profile | At inclusion
  Percentages & Frequencies of cardiovascular risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Leila ABID, MD, Study Chair — The Tunisian Society of Cardiology and CardioVascular Surgery
Locations (1):
- The Tunisian Society of Cardiology and CardioVascular Surgery, Tunis, Tunisia

REFERENCES:
- [Derived] Abid L, Hammami R, Abdesselem S, Boudiche S, Hedi BS, Sayahi K, Bahloul A, Chamtouri I, Charfeddine S, Rais L, Drissa M, Ben Kaab B, Ibn Hadj Amor H, Ben Fatma L, Garbaa R, Boukhris S, Emna A, Ben Halima M, Amdouni N, Ghorbel S, Soudani S, Khaled I, Triki S, Bouazizi F, Jemai I, Abdeljalil O, Ammar Y, Farah A, Neji A, Oumaya Z, Seghaier S, Mokrani S, Thawaba H, Sarray H, Ouaghlani K, Thabet H, Mnif Z, Fatma BM, Sghaier M, Khalifa R, Fourati S, Kammoun Y, Abid S, Hamza C, Ben Jeddou S, Sabbah L, Lakhdhar R, Dammak N, Sellami T, Herbegue B, Koubaa A, Triki F, Ellouze T, Hmoudi A, Ben Ameur I, Boukhchina MM, Abid N, Ouechtati W, Nasrallah N, Houidi Y, Mghaieth Zghal F, Elhem G, Chayeb M, Sarra C, Kaabachi S, Saadaoui N, Ben Ameur I, Affes M, Ouali S, Chaker M, Naana H, Meriem D, Jarrar M, Mnif J, Turki A, Zairi I, Langar J, Dardouri S, Hachaichi I, Chettaoui R, Smat W, Chakroun A, Mzoughi K, Mechmeche R, Ben Halima A, Ben Kahla Koubaa S, Chtourou S, Mohamed Abdelkader M, Ayari M, Hadrich M, Rami T, Azaiez F, Bouhlel I, Sahnoun S, Jerbi H, Imtinene BM, Riahi L, Sahnoun M, Ben Jemaa A, Ben Salem A, Rekik B, Ben Doudou M, Boujnah MR, Joulak A, Omar A, Razgallah R, Sami M, Neffati E, Gamra H, Ben Youssef S, Sdiri W, Ben Halima N, Ben Ameur Y, Kachboura S, Kraiem S, Fehri W, Zakhama L, Bezdah L, Mohamed Sami M, Drissa H, Maatouk MF, Kammoun S, Addad F. Design and Rationale of the National Observational Multicentric Tunisian Registry of Hypertension: Protocol for Evaluating Hypertensive Patient Care in Clinical Practice. JMIR Res Protoc. 2022 Sep 2;11(9):e21878. doi: 10.2196/21878. PMID 36053572
- See also: STCCCV website — http://www.stcccv.org.tn/
- See also: STCCCV FaceBook page — http://www.facebook.com/Soci%C3%A9t%C3%A9-Tunisienne-de-Cardiologie-et-de-Chirurgie-Cardio-Vasculaire-158326807565380/
- See also: https://journals.lww.com/jhypertension/Abstract/2021/04001/IMPACT_OF_OVERWEIGHT_AND_OBESITY_ON_BLOOD_PRESSURE.1022.aspx — https://journals.lww.com/jhypertension/Abstract/2021/04001/IMPACT_OF_OVERWEIGHT_AND_OBESITY_ON_BLOOD_PRESSURE.1022.aspx
- See also: HYPERTENSION MANAGEMENT DURING RAMADAN: RESULTS FROM THE NATIONAL TUNISIAN REGISTRY OF HYPERTENSION (NATURE HTN) — https://journals.lww.com/jhypertension/Abstract/2021/04001/HYPERTENSION_MANAGEMENT_DURING_RAMADAN__RESULTS.414.aspx
- See also: BLOOD PRESSURE CONTROL OF HYPERTENSIVE PATIENTS WITH HIGH HEART RATE (RESULTS FROM NATURE HTN) — https://journals.lww.com/jhypertension/Abstract/2021/04001/BLOOD_PRESSURE_CONTROL_OF_HYPERTENSIVE_PATIENTS.833.aspx
- See also: Epidemiologic features and management of hypertension in Tunisia, the results from the Hypertension National Registry (NaTuRe HTN) — https://bmccardiovascdisord.biomedcentral.com/articles/10.1186/s12872-022-02584-y?fbclid=IwAR0NnoP1GM51dxD1gmLVsrETUg0mDj0_Wtp4hDoDIZkRMQswt54_t18Lq7c